CLINICAL TRIAL: NCT01710423
Title: Improving Home Food Preparation Practices Among Families With Young Children: A Peer Mentoring Intervention
Brief Title: Peer-mentored Cooking Classes for Parents of Toddlers: Do Families Cook More and Eat Healthier After the Intervention?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-009579
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
Keywords: Obesity; Nutrition; Home Food Preparation; Peer Mentoring; Early Head Start; Cooking; Diet
MeSH Terms: conditions — Obesity | interventions — Cooking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Intervention (Experimental): Peer mentoring intervention ('Cooking with Friends')
  Interventions: Behavioral: Peer mentoring intervention ('Cooking with Friends')
- Delayed Entry Control (No Intervention)

INTERVENTIONS:
Behavioral: Peer mentoring intervention ('Cooking with Friends') — 'Cooking with Friends' is a community-located, peer mentoring intervention aimed at improving home food preparation practices in families with young children.
  The intervention was developed in an iterative, community-based research approach, and will be conducted in partnership with Early Head Start (EHS) at The Children's Hospital of Philadelphia. Cooking with Friends builds on existing monthly cooking classes at EHS that have proven popular with EHS families. Through 5 weekly classes, this intervention will explore topics of how to prepare healthy foods at home.
  The peer mentoring component is a novel innovation to this intervention. The intervention pairs peer mentors to individual mentees in a community setting, to effect behavioral change among caregivers of young children.
  Arms: Immediate Intervention

SUMMARY:
This study aims to test the effectiveness of a community-located, peer mentored intervention to improve home food preparation practices in families with young children.

DETAILED DESCRIPTION:
Barriers to healthy eating and active living are at the heart of the obesity epidemic. This study focuses on a key factor underlying healthy eating: home food preparation. Preparing food at home entails a sequence of steps from obtaining food, to planning and cooking or preparing meals, to finally serving and eating the meal. Many strategies to curb obesity in children focus on eliminating processed and fast food from the diet, as well as improving access to fresh produce and other healthy ingredients. A collective ability to regularly and reliably prepare healthy food at home is implicit in these and other prevention strategies. Little research, however, has grappled with the phenomenon that there has been a generational loss of home food preparation ability over the past few decades. What is urgently needed is to design effective, enticing, and scalable interventions to improve home food preparation practices across diverse groups.

This study aims to test the effectiveness of a community-located, peer mentored intervention to improve home food preparation practices in families with young children. The investigators will partner with Children's Hospital of Philadelphia Early Head Start, a community-based organization serving families with children ages 0 to 3 years in West Philadelphia, aiming specifically to:

1. Use the principles of Community Based Participatory Research (CBPR) to design, evaluate and disseminate a peer mentored intervention aimed at improving home food preparation practices among families with young children.
2. Conduct a randomized controlled trial with a delayed entry control group to test the effect of the intervention on three outcomes: home food preparation practices, healthfulness of the diet, and cooking-related self-efficacy.

The investigators hypothesize that families participating in this intervention will demonstrate improvement in parental self-efficacy related to cooking, home food preparation practices, and the healthfulness of parents' and toddlers' diets post-intervention, compared to families who do not participate in the intervention.

ELIGIBILITY:
Mentee Inclusion Criteria:

1. Eligible mentees will be caregivers of 0-3 year old children who are enrolled in Early Head Start at The Children's Hospital of Philadelphia (CHOP EHS) at the time of recruitment.
2. Caregiver enrollment in CHOP EHS requires the following:

   1. Children are 0-3 years old (Expectant mothers are also eligible to enroll)
   2. The family has an income at or below federal poverty level
   3. The family lives in West Philadelphia, within the geographic area served by CHOP EHS.
3. Caregiver is able to give informed consent.

Mentor Inclusion Criteria:

1. Eligible peer mentors should meet the inclusion criteria set for above for mentees.
2. The study team, in conjunction with EHS staff, will decide which participants will be invited to be peer mentors, based on attributes including interest, leadership ability, and home food preparation skills.

Children Inclusion Criteria:

1. 0-3 year old children of mentee caregivers enrolled in the study
2. If a mentee caregiver has more than one child currently enrolled in CHOP EHS, then all their eligible children will be enrolled in the study.
3. If there are expectant mothers who are enrolled as mentees, their children will be enrolled in the study upon delivery.

Exclusion Criteria:

1. Caregivers and children not meeting the inclusion criteria above.
2. Subjects who, in the opinion of the Investigator, may be unable to participate in the study schedules or procedures.
3. Children of peer mentors will not be eligible for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Food Frequency Questionnaire | 23 weeks from Baseline
  The primary outcome will be the change in healthfulness of the diet as measured by food frequency questionnaires for participants through the course of the study. Study staff will meet with each participant and ask them to answer questions about the frequency of their food and beverage consumption over the course of a 12 month period. The results will be analyzed for consumption of specific food-groups (fruits, vegetables, whole grains, dairy, etc.). The primary endpoint is the difference in the healthfulness of the diet between the immediate intervention group and the control group at week 23.

SECONDARY OUTCOMES:
Cooking-related self-efficacy | 23 weeks from Baseline
  Self-efficacy related to cooking will be measured using a 25-item instrument. We will assess to assess the difference between the immediate intervention group and the control group at week 23.
Home food preparation practices | 23 weeks from Baseline
  Home food preparation practices will be measured using questions from the National Health and Nutrition Examination Survey. We will measure the difference in home food preparation practices between the immediate intervention group and the control group at week 23.
Body mass index | 41 weeks from Baseline
  We will measure the change in parent and child body mass index before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Senbagam Virudachalam, MD, MSHP, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States